CLINICAL TRIAL: NCT03286699
Title: Leukocyte Telomere Length: Diet and Exercise Trial
Brief Title: Lifestyle Change for Better Health
Acronym: LCBH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to challenges with recruitment, we were unable to complete recruitment as planned during the period we had funding to do so.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dana Bovbjerg, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY19070303; R21CA212628 (NIH)
Record Dates: First submitted 2017-01-31; First posted 2017-09-18 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer; Telomere Shortening; Colorectal Adenoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DIET (Active Comparator): This group will be prescribed a Dietary Intervention that reduces energy intake by 500-1000 kcal/day and induces a weight loss of approximately 1-2 pounds per week during the intervention, with the weight loss goal individualized to each participant.
  Interventions: Behavioral: Dietary Intervention
- DIET-PA (Active Comparator): This group will be prescribed a Dietary Intervention that reduces energy intake by 500-1000 kcal/day and induces a weight loss of approximately 1-2 pounds per week during the intervention, with the weight loss goal individualized to each participant. In addition, this group will be prescribed moderate-intensity Physical Activity Intervention that will progressively increase to the goal of 250 minutes/week.
  Interventions: Behavioral: Dietary Intervention; Behavioral: Physical Activity Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — The behavioral weight loss intervention strategies will not be limited to, self-monitoring, goal setting, problem solving, mastery skills, social support, and relapse prevention. Participants will receive a standard behavioral weight control program, delivered on a one-on-one basis. They will attend in-person sessions (~30-45 minutes) with time to: distribute intervention materials, interact with the participant, identify participants that need additional support, and conduct the intervention. Each in-person visit focuses on a specific behavioral topic related to weight loss to address eating behaviors. Subjects will also participate in phone calls with the interventionist (~10 minutes). Depending on the week, subjects will have between 10 and 45 minutes of total intervention contact.
Behavioral: Physical Activity Intervention — The behavioral weight loss intervention strategies will not be limited to, self-monitoring, goal setting, problem solving, mastery skills, social support, and relapse prevention. Participants will receive a standard behavioral weight control program, delivered on a one-on-one basis. They will attend in-person sessions (~30-45 minutes) with time to: distribute intervention materials, interact with the participant, identify participants that need additional support, and conduct the intervention. Each in-person visit focuses on a specific behavioral topic related to weight loss to address physical activity behaviors. Subjects will also participate in phone calls with the interventionist (~10 minutes). Depending on the week, subjects will have 10 to 45 minutes of total intervention contact.
  Arms: DIET-PA

SUMMARY:
The goal of the research is to provide a first critical test of the novel scientific idea that a combined diet and exercise intervention may ameliorate shortening of leukocyte telomere length (LTL) in individuals with histories of successfully treated non-metastatic bladder cancer (BC) or colorectal adenoma (CRA) compared to a diet only intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25.0 to <40 kg/m2 (allows for use of assessments such as DXA to be included)
* History of histologically confirmed bladder cancer (non-metastatic) or colorectal adenoma
* Under clinical surveillance with no evidence of disease

Exclusion Criteria:

* WHO performance status 3-4 or deemed physically unable to participate by physician
* Currently pregnant or breastfeeding, were pregnant in the previous 6 months or breastfeeding in the previous 3 months, or planning pregnancy in the next year
* History of bariatric surgery
* Medical condition that could affect body weight (e.g., diabetes mellitus, hyperthyroidism, uncontrolled hypothyroidism, chronic renal insufficiency, chronic liver disease, gastrointestinal disorders including ulcerative colitis)
* Cancer diagnosis (other than bladder cancer or non-melanoma skin cancer) in the previous 5 years
* Current congestive heart failure, signs or symptoms indicative of an increased acute risk for a cardiovascular event
* History of myocardial infarction, coronary artery bypass or angioplasty, conditions requiring chronic anticoagulation (recent or recurrent DVT)
* Resting systolic blood pressure of >160 mmHg or diastolic blood pressure >100 mmHg
* Eating disorder that would contraindicate weight loss or physical activity
* Alcohol or substance abuse
* Current treatment for psychiatric issues (e.g., depression, bipolar disorder) or taking daily or extended release psychotropic medications in the previous 12 months
* Report exercising more than 100 minutes per week over the past 3 months (NOTE: includes physical activity performed for sport, fitness, or recreational activity; physical activity performed as part of occupation or household chores is not included)
* Weight loss of greater than 5% or participating in a weight reduction diet in the past 3 months
* Report plans to relocate to a location not accessible to the study site or having employment, personal, or travel commitments that prohibit attendance to at least 80 percent of the scheduled intervention sessions and all of the scheduled assessments

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Leukocyte telomere length (LTL) at the 6 month assessment (controlling for appropriate covariates) | Blood samples will be collected as part of the 6 month assessment
  LTL will be measured in blood samples from participants

SECONDARY OUTCOMES:
Leukocyte telomere length (LTL) at the 3 month assessment (controlling for appropriate covariates) | Blood samples will be collected as part of the 3 month assessment
  LTL will be measured in blood samples from participants
Leukocyte telomere length (LTL) at the 12 month assessment (controlling for appropriate covariates) | Blood samples will be collected as part of the 12 month assessment (as feasible)
  LTL will be measured in blood samples from participants
Telomerase level at 3 months (controlling for appropriate covariates) | Blood samples will be collected as part of the 3 month assessment
  Telomerase will be measured in blood samples from participants
Telomerase level at 6 months (controlling for appropriate covariates) | Blood samples will be collected as part of the 6 month assessment
  Telomerase will be measured in blood samples from participants
Telomerase level at 12 months (controlling for appropriate covariates) | Blood samples will be collected as part of the 12 month assessment (as feasible)
  Telomerase will be measured in blood samples from participants
8-OHdG level at 3 months (controlling for appropriate covariates) | Samples will be collected as part of the 3 month assessment
  8-OHdG will be measured in samples from participants
8-OHdG level at 6 months (controlling for appropriate covariates) | Samples will be collected as part of the 6 month assessment
  8-OHdG will be measured in samples from participants
Superoxide dismutase 1 (SOD1) at 3 months (controlling for appropriate covariates) | Samples will be collected as part of the 3 month assessment
  SOD1 will be measured in samples from participants
Superoxide dismutase 1 (SOD1) at 6 months (controlling for appropriate covariates) | Samples will be collected as part of the 6 month assessment
  SOD1 will be measured in samples from participants
Superoxide dismutase 2 (SOD2) at 3 months (controlling for appropriate covariates) | Samples will be collected as part of the 3 month assessment
  SOD2 will be measured in samples from participants
Superoxide dismutase 2 (SOD2) at 6 months (controlling for appropriate covariates) | Samples will be collected as part of the 6 month assessment
  SOD2 will be measured in samples from participants
Glutathione peroxidase (Gpx) at 3 months (controlling for appropriate covariates) | Samples will be collected as part of the 3 month assessment
  Gpx will be measured in samples from participants
Glutathione peroxidase (Gpx) at 6 months (controlling for appropriate covariates) | Samples will be collected as part of the 6 month assessment
  Gpx will be measured in samples from participants
Systemic Inflammatory Response (SIR) at 3 months (controlling for appropriate covariates) | Samples will be collected as part of the 3 month assessment
  SIR will be measured in samples from participants
Systemic Inflammatory Response (SIR) at 6 months (controlling for appropriate covariates) | Samples will be collected as part of the 6 month assessment
  SIR will be measured in samples from participants

OTHER OUTCOMES:
Body Mass Index (BMI) at 3 months (controlling for appropriate covariates) | Measurements will be collected as part of the 3 month assessment
  BMI will be calculated from height and weight measurements
Body Mass Index (BMI) at 6 months (controlling for appropriate covariates) | Measurements will be collected as part of the 6 month assessment
  BMI will be calculated from height and weight measurements
Body composition at 3 months (controlling for appropriate covariates) | Measurements will be collected as part of the 3 month assessment
  Body composition will be measured by dual-energy x-ray absorptiometry (DXA)
Body composition at 6 months (controlling for appropriate covariates) | Measurements will be collected as part of the 6 month assessment
  Body composition will be measured by dual-energy x-ray absorptiometry (DXA)
Regional adiposity (DXA) at 3 months (controlling for appropriate covariates) | Measurements will be collected as part of the 3 month assessment
  Regional adiposity will be measured by dual-energy x-ray absorptiometry (DXA)
Regional adiposity (DXA) at 6 months (controlling for appropriate covariates) | Measurements will be collected as part of the 6 month assessment
  Regional adiposity will be measured by dual-energy x-ray absorptiometry (DXA)
Waist-to-hip ratio at 3 months (controlling for appropriate covariates) | Measurements will be collected as part of the 3 month assessment
  Waist-to-hip ratio will be calculated from waist and hip measurements
Waist-to-hip ratio at 6 months (controlling for appropriate covariates) | Measurements will be collected as part of the 6 month assessment
  Waist-to-hip ratio will be calculated from waist and hip measurements
Objective physical activity level at 3 months (controlling for appropriate covariates) | Total physical activity will be calculated from measurements collected for 7 consecutive days following the 3 month assessment
  Physical Activity will be objectively measured with SenseWear BodyMedia
Objective physical activity level at 6 months (controlling for appropriate covariates) | Total physical activity will be calculated from measurements collected for 7 consecutive days following the 6 month assessment
  Physical Activity will be objectively measured with SenseWear BodyMedia
Self-reported physical activity level at 3 months (controlling for appropriate covariates) | Self-reports will be obtained as part of the 3 month assessment
  The Paffenbarger Physical Activity Questionnaire will be used to obtain a self-reported measure of physical activity
Self-reported physical activity level at 6 months (controlling for appropriate covariates) | Self-reports will be obtained as part of the 6 month assessment
  The Paffenbarger Physical Activity Questionnaire will be used to obtain a self-reported measure of physical activity
Cardiorespiratory fitness at 3 months (controlling for appropriate covariates) | Measurements will be collected as part of the 3 month assessment
  Cardiorespiratory Fitness (oxygen consumption) will be measured by submaximal treadmill test
Cardiorespiratory fitness at 6 months (controlling for appropriate covariates) | Measurements will be collected as part of the 6 month assessment
  Cardiorespiratory Fitness (oxygen consumption) will be measured by submaximal treadmill test
Depressive symptoms at 3 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 3 month assessment
  The Center for Epidemiologic Studies Depression Scale will be used to obtain a self-reported measure of depressive symptoms
Depressive symptoms at 6 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 6 month assessment
  The Center for Epidemiologic Studies Depression Scale will be used to obtain a self-reported measure of depressive symptoms
Symptoms of anxiety at 3 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 3 month assessment
  The State subscale of the State Trait Anxiety Inventory will be used to obtain a self-reported measure of acute anxiety
Symptoms of anxiety at 6 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 6 month assessment
  The State subscale of the State Trait Anxiety Inventory will be used to obtain a self-reported measure of acute anxiety
Perceived stress at 3 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 3 month assessment
  The Perceived Stress Scale will be used to obtain a self-reported measure of perceived stress
Perceived stress at 6 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 6 month assessment
  The Perceived Stress Scale will be used to obtain a self-reported measure of perceived stress
Sleep quality at 3 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 3 month assessment
  The Pittsburgh Sleep Quality Index will be used to obtain a self-reported measure of overall sleep quality
Sleep quality at 6 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 6 month assessment
  The Pittsburgh Sleep Quality Index will be used to obtain a self-reported measure of overall sleep quality
Quality of life at 3 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 3 month assessment
  The Functional Assessment of Cancer Therapy - Bladder Cancer will be used to obtain a self-reported measure of health-related quality of life
Quality of life at 6 months (controlling for appropriate covariates) | Questionnaires will be completed as part of the 6 month assessment
  The Functional Assessment of Cancer Therapy - Bladder Cancer will be used to obtain a self-reported measure of health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dana Bovbjerg, PhD, Principal Investigator — University of Pittsburgh; John Jakicic, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No